CLINICAL TRIAL: NCT02062112
Title: Comparison of Patterns of Laxative Ingestion to Improve Bowel Preparation for Colonoscopy: A Pilot Randomized Trial
Brief Title: Improving Tolerability of Bowel Preparation Laxative for Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Howard University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB-13-MED-60
Record Dates: First submitted 2014-02-11; First posted 2014-02-13 (Estimated); Last update posted 2018-09-14 (Actual); Status verified 2018-09

CONDITIONS: Colonoscopy; Bowel Preparation
Keywords: Bowel preparation solutions; Colonoscopy; Polyethylene glycol

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (3):
- Unflavored group (No Intervention): The patient will mix 1 gallon of polyethylene glycol with water and drink as directed by his/her endoscopist. No flavoring will be added.
- Flavored group (Active Comparator): The patient will mix 1 gallon of polyethylene glycol with water, add flavoring to the entire solution and drink at the time specified by his/her endoscopist.
  Interventions: Other: Pattern of flavoring of bowel laxative
- Liberal group (Active Comparator): The patient will mix 1 gallon of polyethylene glycol with water. Fill 2 cups with the solution. The patient will add flavoring to one cup and drink both the flavored and unflavored solutions in the cups. The patient will then determine how he/she wants to drink the rest of the bowel preparation laxatives based on their taste preference and drink at the time specified by his/her endoscopist.
  Interventions: Other: Pattern of flavoring of bowel laxative

INTERVENTIONS:
Other: Pattern of flavoring of bowel laxative — Unflavored bowel laxative versus entire bowel laxative flavored versus liberal flavoring as decided by patient
  Arms: Flavored group; Liberal group

SUMMARY:
The purpose of this study is to determine whether the pattern of flavoring and drinking of laxatives for colonoscopy can improve the experience of patients when they are undergoing bowel preparation for the test.

Investigators hypothesize that patients will have a better experience if patients taste the bowel preparation laxative with and without flavoring and then decide how they want to drink the rest of the laxative since taste preferences vary widely from person to person.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years and older) referred for outpatient colonoscopy

Exclusion Criteria:

* Patients with history of bowel resection
* patients with history of inflammatory bowel disease
* History of polyposis syndrome
* History of colorectal cancer
* History of poor taste perception from any cause

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 313 (Actual)
Dates: Start 2014-02-11 (Actual); Primary Completion 2015-01-21 (Actual); Study Completion 2015-01-21 (Actual)

PRIMARY OUTCOMES:
Overall patients' experience with the bowel preparation process with ratings from 1 (unbearable) to 10 (Pleasant) | At the time of colonoscopy
  On the day of the patient's colonoscopy, each patient will complete another form regarding their bowel preparation experience. Information gathered will include their ratings of the bowel preparation laxative's taste, ease of consumption, presence or absence of nausea, vomiting, whether they consumed the entire recommended laxative and their overall ratings of the bowel preparation experience.

SECONDARY OUTCOMES:
Endoscopist ratings of the patient's bowel preparation quality using Aronchick scale | At the colonoscopy
  During the colonoscopy, the endoscopist who will be masked to the assignment of the patients will assess the quality of bowel preparation and grade as Poor/Inadequate, Fair, Good, Very Good or Excellent.

OTHER OUTCOMES:
Prevalence of colorectal neoplasia (polyps, adenoma and cancer) | At the colonoscopy
  The detection of colorectal lesions during colonoscopy (polyps, adenoma and cancer)
Correlation of beverage intake patterns with tolerability of bowel laxatives | At the time of colonoscopy
  Investigators will examine patients' preferred pattern of non-alcoholic beverage intake for coffee, tea and carbonated drinks with their bowel preparation experience

CONTACTS AND LOCATIONS:
Overall Officials: Adeyinka O Laiyemo, MD, MPH, Principal Investigator — Howard University
Locations (1):
- Howard University, Washington D.C., District of Columbia, United States

REFERENCES:
- [Background] Hayes A, Buffum M, Fuller D. Bowel preparation comparison: flavored versus unflavored colyte. Gastroenterol Nurs. 2003 May-Jun;26(3):106-9. doi: 10.1097/00001610-200305000-00004. PMID 12811320